CLINICAL TRIAL: NCT04535258
Title: Blended Treatment for Alcohol Use Disorder - The BLEND-A Study Evaluation of a Blended Treatment Intervention for Alcohol Use Disorder in Denmark
Brief Title: Blended Treatment for Alcohol Use Disorder
Acronym: BLEND-A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BLEND-A
Record Dates: First submitted 2020-04-24; First posted 2020-09-01 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized (18 institutions, 4 waves)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First-movers (Other): The first four alcohol clinics offers internet-based treatment to the patients who chooses the proportion of internet-based sessions.
  Interventions: Device: Blend-A
- Second-movers (Other): After three months, the next five alcohol clinics offers internet-based treatment to the patients who chooses the proportion of internet-based sessions.
  Interventions: Device: Blend-A
- Third-movers (Other): After three months, the next five alcohol clinics offers internet-based treatment to the patients who chooses the proportion of internet-based sessions.
  Interventions: Device: Blend-A
- Fourth-movers (Other): After three months, the last four alcohol clinics offers internet-based treatment to the patients who chooses the proportion of internet-based sessions.
  Interventions: Device: Blend-A

INTERVENTIONS:
Device: Blend-A — Treatment for alcohol use disorders will be offered also as an internet-based option.

SUMMARY:
Blended Treatment for Alcohol Use Disorder (BLEND-A) is a pragmatic, cluster randomized controlled trial to assess the clinical effectiveness and cost-effectiveness of implementing a blended treatment format that aims to reduce problematic alcohol use. Blended treatment is a treatment format where treatment as usual is offered as a combination of online and face-to-face sessions, integrated into one treatment protocol. The BLEND-A study will evaluate and implement a blended treatment program in routine alcohol addiction treatment. The trial is led by Unit of Clinical Alcohol Research, University of Southern Denmark (UCAR) in collaboration with partners at the Centre for Telepsychiatry in the Region of Southern Denmark (CTP), and Sundhed.dk.

DETAILED DESCRIPTION:
Background: A major challenge to psychological treatment for Alcohol Use Disorder (AUD) is patient non-compliance. A promising new treatment approach that is hypothesized to increase treatment compliance is blended treatment, consisting of face-to-face contact with a therapist combined with modules delivered over the Internet within the same protocol. While this treatment concept has been developed and proven effective for a variety of mental disorders, it has not yet been examined for AUD.

Aims: The study described in this protocol aims to examine and evaluate patient compliance with blended AUD treatment as well as the clinical and cost effectiveness of such treatment compared to face-to-face treatment only.

Methods: The study design is a pragmatic, stepped-wedge cluster randomized controlled trial. The included outpatient institutions (planned number of patients: n=1800) will be randomized in clusters to implement either blended AUD treatment or face-to-face treatment only, i.e. treatment as usual (TAU). Both treatment approaches consist of motivational interviewing and cognitive behavioral therapy. Data on socio-demographics, alcohol consumption, addiction severity, treatment retention, treatment duration and intensity, and type of conclusion of treatment (dropout vs. compliance), will be retrieved from the National Register of Alcohol Treatment (NAB). In addition, all patients will be assessed for alcohol consumption, consequences of drinking and quality of life at treatment entry and six months after treatment conclusion. Data will be analyzed with an Intention-to-treat approach by means of generalized mixed models with random effect for cluster and fixed effect for each step. Also, analyses evaluating cost-effectiveness will be conducted.

Discussion: Blended treatment may increase treatment compliance and thus improve treatment outcomes due to increased flexibility of the treatment course. Since this study is conducted within an implementation framework it can easily be scaled up, and blended treatment has the potential to become an alternative offer in the majority ofmany outpatient clinics nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Legal person seeking public alcohol treatment in the participating municipalities.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance and premature dropout in alcohol treatment | One year after enrolled in the study
  BLEND-A (outpatient treatment as usual offered as a combination between face-to face and internet-based sessions) leads to a change in compliance in treatment during one year following initiation of treatment, compared to TAU (usual treatment delivered as face-to-face outpatient treatment only ), and measured as a change in premature dropout of treatment in the National Register of alcohol treatment (NAB).
Effectiveness of alcohol treatment | 6 months after enrolled in the study
  The effectiveness of BLEND-A compared to TAU, measured by alcohol intake 6 months after treatment start. The alcohol intake is measured by self-reported alcohol intake.

SECONDARY OUTCOMES:
Differences in Quality of Life according to the intervention | 6 months after enrolled in the study
  BLEND-A leads to a change in quality of life (measured by means of Patient Reported Outcomes (PRO)) among patients, compared to face-to-face outpatient treatment as usual, measured 6 months after treatment start.
Which part of treatment is appreciated to receive via the internet | Through study completion, an average of 1 year
  Based on the user data from BLEND-A, we expect to be able to determine what part of the usual treatment that is appreciated to receive via the internet.
Optimal blend | Through study completion, an average of 1 year
  Based on the user data from BLEND-A, we expect to be able to determine the optimal combination of face-to-face and internet-based sessions.

OTHER OUTCOMES:
Qualitative interviews | Through study completion, an average of 1 year
  The perspectives for further refinement of BLEND-A will be assessed by qualitative interviews with patients and therapists receiving or delivering the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anette S. Nielsen, PhD, Study Director — University of Southern Denmark
Locations (1):
- Unit if Clinical Alcohol Research, Odense, Denmark

REFERENCES:
- [Derived] Tarp K, Christiansen R, Bilberg R, Borkner S, Dalsgaard C, Paldam Folker M, Sogaard Nielsen A. Patient Perspectives on Blended Internet-Based and Face-to-Face Cognitive Behavioral Therapy for Alcohol Use Disorder: Qualitative Study. J Med Internet Res. 2024 Oct 23;26:e47083. doi: 10.2196/47083. PMID 39441642
- [Derived] Mellentin AI, Behrendt S, Bilberg R, Blankers M, Folker MP, Tarp K, Uffelmann J, Nielsen AS. BLEND-A: blending internet treatment into conventional face-to-face treatment for alcohol use disorder - a study protocol. BMC Psychiatry. 2021 Mar 6;21(1):131. doi: 10.1186/s12888-021-03122-4. PMID 33676429